CLINICAL TRIAL: NCT00585104
Title: Myocardial Hemodynamic Effects of Levosimendan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19266; IRB# 00019266
Record Dates: First submitted 2007-12-21; First posted 2008-01-03 (Estimated); Results first posted 2010-06-09 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Simendan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): All randomized patients receive drug.
  Interventions: Drug: levosimendan

INTERVENTIONS:
Drug: levosimendan — 10-minute infusion
  Other Names: Simdax

SUMMARY:
This study will test the hypothesis that mechanical efficiency as measured by pressure-volume loop assessment should improve during short-term treatment with intravenous levosimendan.

Levosimendan (SimdaxTM, Abbott Laboratories, Abbott Park, IL) is a calcium sensitizer which has been shown to have beneficial hemodynamic effects in patients with decompensated congestive heart failure (CHF). Levosimendan is a new calcium sensitizer that binds to troponin C. This agent is approved in Europe for treatment of heart failure patients. In the United States, this agent is currently under phase III investigation for intravenous treatment of patients with acutely decompensated HF who have dyspnea at rest or with minimal activity. Levosimendan has been studied in these patients with acute HF and is considered experimental in the United States for this population.

ELIGIBILITY:
Inclusion Criteria:

* All patients will have either a sinus or paced atrial rhythm with atrioventricular synchrony on electrocardiography
* All patients will have a history of heart failure diagnosed clinically with history of prior symptoms or signs of heart failure with at least one of the following symptoms within the past month: dyspnea on exertion, orthopnea, paroxysmal nocturnal dyspnea, pedal edema
* In asymptomatic patients, patients may be enrolled if they have at least one of the following clinical signs of heart failure: left ventricular third and/or fourth heart sound, jugular venous pressure >7 mmHg, sustained left ventricular impulse, or pulmonary congestion on auscultation
* all patients will have echocardiographic evidence of left ventricular dysfunction

Exclusion Criteria:

* Under age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Michaels, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Levosimendan, Compare Heart Function and Metabolism: All patients received Levosimendan (12mcg/kg IV bolus over 10 minutes, Abbott Laboratories, Abbott Park, IL). All study measurements occur at baseline and 30-minutes after the initiation of levosimendan.
Period: Overall Study
Arm/Group | Levosimendan, Compare Heart Function and Metabolism
Started | 10
Completed | 6
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Levosimendan, Compare Heart Function and Metabolism
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 59 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 10
Left Ventricular End Diastolic Pressure (LVEDP) [Mean (Standard Deviation); unit: mmHg] | 18 (7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricular End-diastolic Pressure (LVEDP) Using Pressure-volume Catheter.
Description: Left ventricular end-diastolic pressure (LVEDP) recorded from CD Leycom ConductNT software analysis.
Time Frame: From baseline to 30-minutes after levosimendan started.
Population: Ten patients were enrolled. Complete data was available in 6 patients. The primary endpoint was change in left ventricular end diastolic pressure (LVEDP) from baseline to 30-minutes after starting levosimendan. An Intent to Treat (ITT) analysis was performed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Levosimendan, Compare Heart Function and Metabolism
Number analyzed (Participants) | 6
mmHg | 5.67 (4.32)

ADVERSE EVENTS:
Arm/Group | Levosimendan, Compare Heart Function and Metabolism
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Of the ten (10) patients enrolled, only 6 patients completed the study protocol for which we collected data. The data is insufficient to provide a formal summary for publication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No